CLINICAL TRIAL: NCT04434547
Title: A Randomized Controlled Trial on the Effect of Adding Platelets Rich Plasma Intrauterine on the Day of Ovum Pickup in ICSI Patients With Recurrent Implantation Failure
Brief Title: A RCT on the Effect of Platelets Rich Plasma in ICSI Patients With Recurrent Implantation Failure
Acronym: PRP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Osman Hospital (Other)
Responsible Party: Principal Investigator, Dr Hisham Gouda, Assistant prof OB/GYN Cairo university, Dr. Osman Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DrHGouda
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy Outcome
Keywords: PRP , IVF

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): In the PRP group autologous platelets rich plasma was prepared from the blood using the two step centifuge process .Under ultrasound guidance and complete aseptic procedure , 1 ml of PRP was infused inside the uterus while performing the mock embryo transfer
  Interventions: Biological: PRP
- Control group (No Intervention): In the control group mock embryo transfer was performed without injecting anything inside the uterus.

INTERVENTIONS:
Biological: PRP — During the mock embryo transfer on oocyte retrieval day, 1ml of PRP was infused inside the uterus
  Other Names: Platelets rich plasma
  Arms: PRP group

SUMMARY:
This randomized controlled trial will be performed on 86 patients with recurrent implantation failure at Dar El Teb infertility and IVF center . Patients were randomized on a 1 to 1 ratio to platelets rich plasma ( PRP) group and control group.

Ovarian stimulation was achieved using highly purified urinary FSH starting on the 2 nd or 3rd day of the cycle . GnRH agonist ( cetrotide) 0.25 mg SC/ day was administered when the leading follicle reached 14mm in mean diameter and a dose of 10000 IU of HCG was administered when 3 or more follicles were 18mm or more in diameter..

Oocyte retrieval was done under ultrasound guidance and in the PRP group 1 ml of platelets rich plasma was infused inside the uterus while performing the mock embryo transfer while in the control group the mock embryo transfer was performed without injecting anything inside the uterus .

All patients received progesterone supplementation and embryo transfer was performed 3 to 5 days after oocyte retrieval.

BHCG level was done 14 days after Embryo transfer and transvaginal ultrasound was done to confirm pregnancy 4 weeks later.

DETAILED DESCRIPTION:
This two arm, allocation concealed ,assessor blinded randomized controlled trial is to be conducted at Dar ElTeb Infertility and IVF center ,Giza,Egypt between the period between June 2020 and March 2021.

Eighty six patients with recurrent implantation failure were randomized in a 1 to 1 ratio to platelets-rich plasma (PRP) group and the control group . Patients were randomized using computer generated randomization list and sequentially numbered sealed envelopes containing allocation written on a card. The randomization list and the sealed envelopes were prepared by a colleague who is not directly involved in the study . The embryologists and the doctors responsible for follow up of the patients after ovum pickup were blinded to received treatment.

Ovarian stimulation was achieved using highly purified urinary FSH ( HPuFSH) (Fostimon,IBSA, Switzerland) started on the 2nd or 3rd day of menstruation . The initial dose of HPuFSH ranged between 150 and 300 IU/day depending on expected ovarian response. The dose of HPuFSH was modified from stimulation day 5 in steps of 75 units every 2nd or 3rd day depending on serum E2 and follicular development assessed by transvaginal ultrasound.

GnRH agonist ( cetrolix acetate) (cetrotide) 0.25mg SC/day was administered when the leading follicle reached 14 mm in mean diameter and was continued until and including the day of HCG administration .

A dose of 10000 IU of HCG was administered when 3 or more follicles were 18mm or more in mean diameter .

Oocyte retrieval under transvaginal ultrasound guidance was performed 34 hours after HCG administration .

In PRP group autologous platelets rich plasma was prepared from the blood using the two step centrifuge process. Under ultrasound guidance and complete aseptic procedures ,the endometrial thickness was measured then 1 ml of PRP was infused inside the uterus while performing the mock embryo transfer . In the control group mock embryo transfer was performed without injecting anything inside the uterus .

All the patients received progesterone vaginal pessaries ( prontogest, Marcyryl, Egypt) 400mg twice daily , starting on the day of oocyte retrieval and continuing until 12 weeks gestation or negative pregnancy test.

No more than 3 embryos were transferred under ultrasound guidance 3 to 5 days after oocyte retrieval . B HCG level was detected in blood 14 days after Embryo transfer to confirm pregnancy and transvaginal ultrasound was performed 4 weeks after embryo transfer to confirm clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* patients with history of three or more unsuccessful IVF-ET cycles with at least two good quality embryos transferred and candidates for fresh embryo transfer

Exclusion Criteria:

Age less than 18 years or more than 35years and body mass index more than 30 kg/m2.

Patients with PCOS, endometriosis, uterine anomalies , Ashermann syndrome, chronic endometritis, chromosomal abnormalities, increased peripheral NK cells, hereditary thrombophylia and anti phospholipid syndrome

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-10-15 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | Four weeks post intervention
  The presence of a gestational sac by transvaginal ultrasound

SECONDARY OUTCOMES:
Implantation rate | Four weeks post intervention
  The number of gestational sacs detected by ultrasound divided by the number of embryos
Ongoing pregnancy rate | Five months post intervention
  Pregnancies continuing beyond the 20th week
Abortion rate | Five months post intervention
  Pregnancies terminated before 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Gouda, MD, Principal Investigator — Assistant prof Cairo university

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nazari L, Salehpour S, Hosseini MS, Hashemi Moghanjoughi P. The effects of autologous platelet-rich plasma in repeated implantation failure: a randomized controlled trial. Hum Fertil (Camb). 2020 Sep;23(3):209-213. doi: 10.1080/14647273.2019.1569268. Epub 2019 Feb 4. PMID 30714427